CLINICAL TRIAL: NCT04050891
Title: Comparative Study of Ultrasound Guided Combined Interscalene and Supraclavicular Brachial Plexus Block Versus General Anesthesia for Brachioaxillary Surgery in Renal Failure Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, MD Lecturer of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS/17.08.26
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group GA (general anesthesia) (No Intervention): After pre-oxygenation general anesthesia was induced using 2mg/kg propofol, 1μg/kg of fentanyl. After loss of consciousness 0.5 mg/kg of atracurium was injected. The endotracheal tube (ETT) was placed and inflated. The patient was mechanically ventilated to adjust end tidal CO2 between 35 and 40mmHg, anesthesia was maintained using 1.2 % isoflurane diluted in 3L of 50 % oxygen mixed with air. Increments of fentanyl (0.5 μg/kg ) and atracurium 10 mg were used whenever required and the hemodynamic values were maintained within 20% of the basal values.
  At the end of surgery, residual muscle relaxant was reversed with 50µg/kg neostigmine and 0.02 mg/kg atropine.
- group RA (regional anesthesia) (Active Comparator): received combined supraclavicular and interscalene block.The mixture of anesthetic suolution was prepared by 20 ml isobaric bupivacaine 0.5% plus 10ml lidocaine 2% plus 10ml normal saline, total volume was 40ml which is devided into 25ml for suraclavicular block and 15ml for intersalene block
  Interventions: Device: combined supraclavicular and interscalene block

INTERVENTIONS:
Device: combined supraclavicular and interscalene block — Supraclavicular block An in plane approach, a 22G needle 75mm was advanced from lateral to medial to the corner pocket where the lower trunk commonly lies at this area between the subclavian artery medially, first rib inferiorly and the plexus superiorly then 10ml of the mixture local anesthetic was injected, the remaining volume was injected just above and lateral to the subclavian artery.
  Interscalene block After local anesthetic infiltration of the skin, a 22G needle 75mm was inserted in plane approach from lateral to medial toward the inter-scalene groove between the anterior and middle scalene muscles. The anesthetic mixture 15 ml was injected toward C5, C6 cervical nerve roots aiming to block nerves escaped from supraclavicular nerve block.
  Arms: group RA (regional anesthesia)

SUMMARY:
The aim of this study is to evaluate the efficacy of combined supraclavicular and interscalene brachial plexus block in brachio-axillary surgeries in chronic renal failure as a sole anesthetic technique in comparison to general anesthesia.

DETAILED DESCRIPTION:
This randomized open blinded end-point pilot study was implemented at Mansoura University Hospitals. After acceptance of Institutional Research Board (No: MS/17.08.26), sixty patients of chronic renal failure, The American Society of Anesthesiologists (ASA) III, aged from 20 to 60 years old of either sex and planned for brachioaxillary graft interposition vascular surgery were enrolled.

Patients refusal, have allergy to local anesthetic, neurological, neuromuscular, psychiatric disorders, uncompensated hepatic, respiratory or cardiac disease, uncontrolled seizures, coagulation disorders, infection at the block injection site, body mass index more than 30 were excluded.

Written informed consents were obtained. Patients were classified using closed envelop method into two groups; group (GA) received general anesthesia; group (RA) received combined supraclavicular and interscalene block, each group were carried on 30 patients.

All patients were subjected to the preoperative assessment including history taking, clinical examination and assessment of ASA score. All patients subjected to dialysis session one day before the surgery. Basal laboratory investigation as complete blood count, coagulation profile (prothrombin time, international normalized ratio and activated partial thromboplastin time), arterial blood gases, Electrocardiography and echocardiography were done after dialysis.

After an overnight fasting, patients admitted to preanesthetic room where an intravenous (IV) cannula was inserted in the contralateral upper limb. Standard monitoring was applied to the patient include heart rate (HR), noninvasive blood pressure (NIBP), peripheral oxygen saturation (SpO2).

Numerical rating scale (NRS) was explained to all candidates (zero = no pain and 10 = the worst pain). Patients were lightly sedated by fentanyl 0.5 μg /kg IV to maintain verbal contact.

Group (GA):

After pre-oxygenation general anesthesia was induced using 2mg/kg propofol, 1μg/kg of fentanyl. After loss of consciousness 0.5 mg/kg of atracurium was injected. The endotracheal tube (ETT) was placed and inflated. The patient was mechanically ventilated to adjust end tidal CO2 between 35 and 40mmHg, anesthesia was maintained using 1.2 % isoflurane diluted in 3L of 50 % oxygen mixed with air. Increments of fentanyl (0.5 μg/kg ) and atracurium 10 mg were used whenever required and the hemodynamic values were maintained within 20% of the basal values.

At the end of surgery, residual muscle relaxant was reversed with 50µg/kg neostigmine and 0.02 mg/kg atropine. Patients were discharged from post anesthesia care unit according to modified Aldrete recovery score ≥ 9 . Side effects or complications were recorded.

Group (RA):

Equipment Sterile gloves, Sterile gauze, Alcohol and betadine solution for sterilization, 22 gauge 90mm stimulating needle, 3 ml syringe filled with 3ml 2% lidocaine for local infiltration at the site of needle entry, 50 ml syringe filled with local anesthetic prepared for injection, Ultrasound device (philips, clearvue 350,USA) and high frequency (4-12MHZ) Linear probe was used in this study, its depth setting was 2-4cm .

The mixture of anesthetic solution was prepared by 20 ml isobaric bupivacaine 0.5% plus 10ml lidocaine 2% plus 10ml normal saline, total volume was 40ml which is divided into 25ml for supraclavicular block and 15ml for interscalene block .

Patient position The patient was placed in supine position with the head turned 45 degrees to the contralateral side.

Supraclavicular block :

Land marks Subclavian artery pulsation which appears as a pulsatile hypoechoic circle, The nerves appear as multiple hypoechoic circles, the most common appearance is a grape like clusters of 4-6 circles likely resembling the divisions or as vertical line of 3 circles likely representing the trunks of the brachial plexus. First rib which appears as hyperechoic linear line. The pleura can also be visualized as hyperechoic line.

After skin preparation and local anesthetic infiltration of the skin, supraclavicular fossa was scanned to locate the landmarks. If there was difficulty in finding the subclavian artery, the transducer was slide medially to identify the distal carotid artery firstly , then moved laterally to image the subclavian artery which rested on the first rib, the pulsation was confirmed by doppler colour. The nerves will appear just lateral and superior to the artery.

An in plane approach, a 22 gauge needle 75mm was advanced from lateral to medial to the corner pocket where the lower trunk commonly lies at this area between the subclavian artery medially, first rib inferior and the plexus superior then 10ml of the mixture local anesthetic was injected, the remaining volume was injected just above and lateral to the subclavian artery.

Interscalene block Land marks The linear probe was placed at the level of the cricoids cartilage. Carotid artery, anterior scalene muscle, middle scalene muscle, sternomastoid muscle, internal jugular vein and nerves in the inter-scalene groove appear hypoechoic distinctly round or oval were seen.

After local anesthetic infiltration of the skin, a 22 gauge needle 75mm was inserted in plane approach from lateral to medial toward the inter-scalene groove between the anterior and middle scalene muscles. The anesthetic mixture 15 ml was injected toward C5, C6 cervical nerve roots aiming to block nerves escaped from supraclavicular nerve block .

The sensory block will be assessed by pinprick test and recorded in two stages: 0= normal sensation; 1= no pain. Onset of sensory block is the time between the end of injection and total abolition of pinprick sensation. Sensory loss was assessed every 3 minutes until 30 minutes after block. The block was defined as complete when loss of sensation is observed in all tested areas .

Motor loss was assessed every 3 minutes until 30 minutes after injection. The block was defined as complete when loss of movement is observed in all tested areas. Motor block was evaluated in the following stages: 0= no weakness; 1= paresis; 2= paralysis. Onset of motor block is the time gaped between the end of injection to complete motor block .

The onset of surgical anesthesia is defined as the time of loss of pinprick sensation at the skin dermatomes involved in the surgical field and inability to do motor functions specific to each nerve.

After operation, patients transferred to the recovery room and monitored. Heart rate, mean arterial blood pressure and SpO2 were recorded for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* sixty patients of chronic renal failure,
* ASA III,
* aged from 20 to 60 years old
* of either sex
* planned for brachioaxillary graft interposition vascular surgery were enrolled.

Exclusion Criteria:

* Patients refusal,
* have allergy to local anesthetic,
* neurological, neuromuscular, psychiatric disorders,
* uncompensated hepatic, respiratory or cardiac disease,
* uncontrolled seizures,
* coagulation disorders,
* infection at the block injection site,
* body mass index more than 30

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Pain assessment by numerical rating scale | 24 hours after surgery
  was explained to all candidates (zero = no pain and 10 = the worst pain)
satisfaction of the surgeon to the combined block supraclavicular and interscalene during operation | 3 hours
  by VAS from 0 to 100 as 0 represents unsatisfied and 100 represents satisfied
satisfaction of the patients to the combined block | 3 hours
  by VAS from 0 to 100 as 0 represents unsatisfied and 100 represents satisfied
graft potency | up to one month after surgery
  by doppler

SECONDARY OUTCOMES:
The onset and duration of sensory and motor block | 30 minutes after block
  recorded after performing regional block for group (RA) over the whole upper limb.
time to first intravenous analgesic requirement | 24 hours after surgery
  1ug/kg fentanyl was given if NRS ≥4
Number of times of needed analgesia | 24 hours after surgery
  Number of times patients need analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Nevert adel, Al Mansurah, Egypt